CLINICAL TRIAL: NCT05843643
Title: SELECT-SLE: A Phase 3 Program to Evaluate the Safety and Efficacy of Upadacitinib in Subjects With Moderately to Severely Active SLE
Brief Title: Program to Assess Adverse Events and Change in Disease Activity of Oral Upadacitinib in Adult Participants With Moderate to Severe Systemic Lupus Erythematosus
Acronym: SELECT-SLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-699; 2023-503655-10-00 (Other: EU CT)
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE; Upadacitinib; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Study 1- Upadacitinib Dose A (Experimental): Participants will receive upadacitinib dose A once daily for 52 weeks.
  Interventions: Drug: Upadacitinib
- Study 1- Placebo (Placebo Comparator): Participants will receive upadacitinib matching placebo once daily for 52 weeks.
  Interventions: Drug: Placebo
- Study 2- Upadacitinib Dose A (Experimental): Participants will receive upadacitinib dose A once daily for 52 weeks.
  Interventions: Drug: Upadacitinib
- Study 2- Placebo (Placebo Comparator): Participants will receive upadacitinib matching placebo once daily for 52 weeks.
  Interventions: Drug: Placebo
- Study 3- Low Disease Activity Upadacitinib (LDA) Dose A (Experimental): Participants in the upadacitinib arms from Study 1 or Study 2 with LDA will receive upadacitinib dose A once daily for 52 weeks.
  Interventions: Drug: Upadacitinib
- Study 3- Low Disease Activity Upadacitinib Dose B (Experimental): Participants in the upadacitinib arms from Study 1 or Study 2 with LDA will receive upadacitinib dose B once daily for 52 weeks.
  Interventions: Drug: Upadacitinib
- Study 3- No LDA Upadacitinib Dose A (Experimental): Participants in the upadacitinib arms from Study 1 or Study 2 with no LDA will receive upadacitinib dose A once daily for 52 weeks.
  Interventions: Drug: Upadacitinib
- Study 3- Upadacitininb Dose A (Experimental): Participants in the placebo arms of Study 1 or Study 2 will receive upadacitinib Dose A once daily for 52 weeks.
  Interventions: Drug: Upadacitinib
- Study 3- Open Label Upadacitinib Dose A (Experimental): Participants who experience a suspected systemic lupus erythematosus (SLE) flare may receive open label upadacitinib Dose A once daily for the remainder of the study.
  Interventions: Drug: Upadacitinib
- Study 3- Open Label Upadacitinib Dose B (Experimental): Participants who reach >= 65 years of age and are still on study drug may receive open-label upadacitinib Dose B once daily, and participants who experience a suspected SLE flare while on upadacitinib Dose B may receive upadacitinib Dose A for the remainder of the study.
  Interventions: Drug: Upadacitinib
- Study 4- Upadacitinib Dose A (Experimental): Participants receiving upadacitinib Dose A in Study 3 will continue on this dose once daily for 104 weeks.
  Interventions: Drug: Upadacitinib
- Study 4- Upadacitinib Dose B (Experimental): Participants receiving upadacitinib Dose B in Study 3 will continue on this dose once daily for 104 weeks.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablets
  Other Names: RINVOQ
  Arms: Study 1- Upadacitinib Dose A; Study 2- Upadacitinib Dose A; Study 3- Low Disease Activity Upadacitinib (LDA) Dose A; Study 3- Low Disease Activity Upadacitinib Dose B; Study 3- No LDA Upadacitinib Dose A; Study 3- Open Label Upadacitinib Dose A; Study 3- Open Label Upadacitinib Dose B; Study 3- Upadacitininb Dose A; Study 4- Upadacitinib Dose A; Study 4- Upadacitinib Dose B
Drug: Placebo — Oral Tablet
  Arms: Study 1- Placebo; Study 2- Placebo

SUMMARY:
Systemic Lupus Erythematosus (SLE) is an immune-mediated disease associated with inflammation of multiple organ systems. This study will assess how safe and effective upadacitinib is in treating adult participants with moderately to severely active SLE. Adverse events and change in the disease activity will be assessed.

Upadacitinib is an approved drug for rheumatoid arthritis, psoriatic arthritis, and axial spondylarthritis and is being developed for the treatment of SLE. This study is "double-blinded", which means that neither the trial participants nor the study doctors will know who will be given upadacitinib and who will be given placebo (does not contain treatment drug) . This study comprised of 4 sub studies. In Study 1 and Study 2, study doctors put the participants in 1 of the 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to placebo. Eligible participants from Study 1 and Study 2 will enter Study 3 at week 52 to receive specific doses of upadacitinib. Study 4 is a 104-week continued extension if participation is likely to provide a benefit to their SLE. Approximately 500 participants diagnosed with SLE will be enrolled in each of the Study 1 and Study 2 in approximately 320 sites across the world.

Participants will receive oral tablets of upadacitinib or matching placebo once daily for 52 weeks in Study 1 and Study 2. Eligible participants from Study 1 and Study 2 will receive oral tablets of upadacitinib once daily for 52 weeks in Study 3.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of systemic lupus erythematosus (SLE) at least 24 weeks prior to screening as defined by the 2019 European Alliance of Associations for Rheumatology (EULAR)/ American College of Rheumatology (ACR) classification criteria for SLE.
* At Screening, must have at least one of the following:

  * antinuclear antibody (ANA) positive (titer >= 1:80)
  * anti-double stranded deoxyribonucleic acid (dsDNA) positive
  * anti-Smith positive
* Hybrid systemic lupus erythematosus disease activity index (hSLEDAI) >= 6, of which >= 4 points are clinical (not based on laboratory criteria), independently reviewed by the MCDR at Screening. Clinical hSLEDAI score (not based on laboratory criteria) must be re-confirmed as >= 4 at the Baseline visit. Lupus headache or organic brain syndrome do not count towards the hSLEDAI points required for eligibility but should be documented on the hSLEDAI if present.
* Physician's Global Assessment (PhGA) >= 1 during screening period.
* On stable background treatment for >= 60 days prior to Baseline (with the exception of oral corticosteroid [OCS], which must be at a stable dose for >=14 days prior to Baseline) with

  * antimalarial(s) [hydroxychloroquine <= 400 mg daily, chloroquine <= 500 mg daily, quinacrine <= 100 mg daily];
  * and/or prednisone (or prednisone-equivalent) (<= 20 mg daily);
  * and/or no more than 1 of the following: azathioprine (<= 150 mg daily), 6-mercaptopurine (<= 150 mg daily), mycophenolate mofetil (<= 2 g daily), mycophenolate sodium <= 1,440 mg/day, leflunomide (<= 20 mg daily), cyclosporine, tacrolimus, voclosporin (<= 23.7 mg twice daily), methotrexate (<= 25 mg weekly), or mizoribine (<= 150 mg daily).

Exclusion Criteria:

* Class III/IV lupus nephritis that was treated with induction therapy within the 6 months prior to Screening.
* Active neuropsychiatric SLE (excluding lupus headache) within the 6 months prior to Screening.
* SLE overlap syndromes including, but not limited to, rheumatoid arthritis, systemic sclerosis, polymyositis, dermatomyositis, or mixed connective tissue disease (Sjögren's syndrome is permitted).
* Antiphospholipid syndrome and prior unprovoked venous or arterial thrombosis who are not on stable and adequate anticoagulation.
* Two or more episodes of herpes zoster, or one or more episodes of disseminated herpes zoster or herpes zoster ophthalmicus.
* History of malignancy, except for successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix.
* Pregnancy, breastfeeding, or considering becoming pregnant during the study.
* Clinically relevant or significant ECG abnormalities at Screening.
* Planned elective surgery that would impact study procedures or assessments through the completion of the Week 52 assessments.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving British Isles Lupus Assessment Group Based Combined Lupus Assessment (BICLA) Response | At Week 52
  BICLA is a composite responder index based on improvement in organ systems without worsening of the overall condition and improvement in disease activity.

SECONDARY OUTCOMES:
Percentage of Flares Participants Experiencing Over Time. | Week 52
  Flare is defined by the Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) Systemic lupus erythematosus disease activity index (SLEDAI) Flare Index (SFI). An index defining Systemic lupus erythematosus (SLE) flares using changes in the Hybrid SLEDAI (hSLEDAI) score, definitions of worsening signs and symptoms, treatment changes, and Physician's Global Assessment of Disease Activity. Flare rate is number of flares per patient-year.
Percentage of Participants Achieving Systemic Lupus Erythematosus Responder Index (SRI) -4 | At Week 52
  SRI is a composite responder index based on improvement in disease activity (number following SRI indicates numerical improvement in hSLEDAI score) without worsening of the overall condition (no worsening in Physician's Global Assessment (PhGA), < 0.3 point increase) or the development of significant disease activity in new organ systems (no new British Isles Lupus Assessment Group [BILAG] A or > 1 new BILAG B).
Percentage of Participants Achieving Lupus Low Disease Activity State (LLDAS) | At Week 52
  LLDAS is a state of low disease activity based on SLEDAI score (hSLEDAI score <= 4 excluding hSLEDAI activity in major organ systems), absence of SLE disease activity in major organ systems and new disease activity, Physician's Global Assessment (PhGA <= 1), and concomitant medication usage.
Time to First Flare per SELENA SLEDAI Flare Index (SFI) | Week 52
  SFI is an index defining SLE flares using changes in the hSLEDAI score, definitions of worsening signs and symptoms, treatment changes, and Physician's Global Assessment of Disease Activity.
Percentage of Participants Achieving Oral Glucocorticoid Dose <=7.5 mg/day Prednisone-Equivalent | From Week 44 to Week 52
  Achievement of oral glucocorticoid dose <=7.5 mg/day prednisone-equivalent among participants taking >= 10 mg/day prednisone-equivalent at baseline.
Percentage of Participants Achieving >= 50% Improvement in Tender or Swollen Joints | Week 52
  Achievement of >= 50% improvement in tender or swollen joints among participants with >= 3 swollen joints and >= 6 total affected joints at Baseline.
Percentage of Participants Achieving >= 50% reduction in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score | Week 52
  CLASI index used to assess cutaneous manifestations of SLE summarizing the activity of the disease. Scores range from 0 to 70, with higher scores indicating more severity. Achievement of >= 50% reduction in CLASI activity score among participants with baseline score >=10.
Change from Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Version 4 | Baseline to Week 52
  The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants. Participants respond to the questions on a scale from 0 (not at all) to 4 (very much). The FACIT-Fatigue score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue.
Change from Baseline in Lupus Pain Numerical Rating Scale (NRS) | At Week 52
  The Lupus Pain-NRS is a single-item questionnaire in which participants are asked to rate their overall pain level due to lupus over the last week. The Lupus Pain-NRS scores range from 0 to 10, with higher scores indicating a higher level of pain.
Change from Baseline in 36-Item Short Form Health Survey (SF-36) Acute Physical Component Summary (PCS) | Baseline to Week 52
  The SF-36v2® Health Survey Acute is a general HRQoL instrument with extensive use in multiple disease states. The instrument comprises 36 total items (questions) targeting a participants's functional health and well-being in 8 dimensions (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Scoring is totaled into a Physical Component Summary and a Mental Component Summary. Higher scores indicate a better state of health.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (369):
- United States (132):
  - AZ Arthritis and Rheumatology /ID# 261848, Chandler, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC - Flagstaff /ID# 254767, Flagstaff, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 252820, Gilbert, Arizona
  - Arizona Arthritis and Rheumatology Research - Glendale Office /ID# 252824, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 261845, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research /ID# 273555, Peoria, Arizona
  - Arizona Arthritis & Rheumatology Associates - East Bell Road /ID# 252831, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 252825, Phoenix, Arizona
  - HonorHealth Rheumatology /ID# 261953, Scottsdale, Arizona
  - Arizona Arthritis & Rheumatology Associates - Tucson /ID# 252828, Tucson, Arizona
  - Arthritis and Rheumatism Associates /ID# 253033, Jonesboro, Arkansas
  - Kaiser Permanente Lakeview Medical Offices /ID# 253906, Anaheim, California
  - David S. Hallegua MD, A Professional Corporation /ID# 253902, Beverly Hills, California
  - Wallace and Lee Center /ID# 275129, Beverly Hills, California
  - Wallace Rheumatic Studies Center, LLC /ID# 252806, Beverly Hills, California
  - Advanced Clinical Research Center, LLC dba TriWest Research Associates /ID# 272870, Chula Vista, California
  - Providence - St. Jude Medical Center /ID# 252822, Fullerton, California
  - Private Practice - Dr. Chandrakant V. Mehta /ID# 275100, Hemet, California
  - Newport Huntington Medical Group /ID# 252827, Huntington Beach, California
  - Moores Cancer Center at UC San Diego /ID# 253903, La Jolla, California
  - Arthritis & Osteo Medical Ctr /ID# 252812, La Palma, California
  - Wagdy Kades, M.D., Inc /ID# 272065, Los Angeles, California
  - Providence St. Johns Health Center /ID# 253905, Santa Monica, California
  - Millennium Clinical Trials /ID# 252817, Thousand Oaks, California
  - Cohen Medical Centers /ID# 268524, Thousand Oaks, California
  - Solace Research /ID# 275198, Tustin, California
  - Upland Rheumatology Center /ID# 268623, Upland, California
  - University of Colorado Hospital /ID# 253184, Aurora, Colorado
  - Denver Arthritis Clinic /ID# 253189, Denver, Colorado
  - Yale University School of Medicine /ID# 254567, New Haven, Connecticut
  - Arthritis and Rheumatic Disease Specialties /ID# 253624, Aventura, Florida
  - HARAC Research Corp. /ID# 254922, Avon Park, Florida
  - Rheumatology Associates of South Florida (RASF) - Clinical Research /ID# 253623, Boca Raton, Florida
  - Mdr Core Network, Inc /Id# 276704, Boynton Beach, Florida
  - Bay Area Arthritis and Osteo /ID# 253597, Brandon, Florida
  - GNP Consultants, dba, GNP Research /ID# 272868, Cooper City, Florida
  - Duplicate_Believe Clinical Trials /ID# 255427, Coral Springs, Florida
  - International Medical Research /ID# 253617, Daytona Beach, Florida
  - Omega Research Debary, LLC /ID# 254939, DeBary, Florida
  - University of Florida /ID# 261984, Gainesville, Florida
  - Finlay Medical Research - Greenacres /ID# 274902, Greenacres City, Florida
  - Evolution Research Center /ID# 272991, Hialeah, Florida
  - Neoclinical Research /ID# 253614, Hialeah, Florida
  - South Florida Rheumatology /ID# 268525, Hollywood, Florida
  - Encore Research Group-Jacksonville Center for Clinical Research /ID# 257272, Jacksonville, Florida
  - UF Health Rheumatology /ID# 255351, Jacksonville, Florida
  - Life Clinical Trials /ID# 253615, Margate, Florida
  - Lakes Research, LLC /ID# 253621, Miami, Florida
  - University of Miami, Division of Rheumatology /ID# 261594, Miami, Florida
  - Ezy Medical Research /ID# 276221, Miami, Florida
  - HMD Research LLC /ID# 253595, Orlando, Florida
  - University of Central Florida /ID# 261112, Orlando, Florida
  - Millennium Research /ID# 253600, Ormond Beach, Florida
  - Vitalia Research /ID# 272642, Palm Beach Gardens, Florida
  - Believe Clinical Trials /ID# 277004, Plant City, Florida
  - IRIS Research and Development, LLC /ID# 253618, Plantation, Florida
  - BayCare Medical Group /ID# 253593, St. Petersburg, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 253602, Tampa, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 253899, Tampa, Florida
  - Baycare Medical Group - Tampa /ID# 255135, Tampa, Florida
  - Emory University School Of Medicine - Atlanta /ID# 261529, Atlanta, Georgia
  - Trinity Research Centers /ID# 262039, Kennesaw, Georgia
  - Atlanta Research Center For Rheumatology - Marietta /ID# 253610, Marietta, Georgia
  - Arthritis and Rheumatology Center PC /ID# 275994, Roswell, Georgia
  - Immunology and Rheumatology Research Associates LLC /ID# 267582, Suwanee, Georgia
  - University of Illinois Hospital and Health Sciences System /ID# 263014, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 264090, Chicago, Illinois
  - Next Innovative Clinical Research - Chicago /ID# 268739, Chicago, Illinois
  - University of Chicago Medical Center /ID# 263162, Chicago, Illinois
  - Deerbrook Medical Associates /ID# 253029, Libertyville, Illinois
  - Illinois Bone & Joint Institute - Morton /ID# 274455, Morton, Illinois
  - Advanced Quality Medical Research /ID# 254983, Orland Park, Illinois
  - OrthoIllinois /ID# 253188, Rockford, Illinois
  - Greater Chicago Specialty Physicians /ID# 253021, Schaumburg, Illinois
  - Clinic Of Dr. Robert Hozman/Clinical Investigation Specialists, Inc /ID# 253020, Skokie, Illinois
  - NorthShore University HealthSystem - Skokie /ID# 254568, Skokie, Illinois
  - Willow Rheumatology and Wellness, PLLC /ID# 253018, Willowbrook, Illinois
  - Western KY Rheumatology /ID# 254937, Hopkinsville, Kentucky
  - Accurate Clinical Research (SMO/Network/Consortium) /ID# 272647, Lake Charles, Louisiana
  - Willis Knighton /ID# 256343, Shreveport, Louisiana
  - University of Maryland, Baltimore /ID# 262556, Baltimore, Maryland
  - UMass Memorial Medical Center /ID# 262742, Worcester, Massachusetts
  - Clinical Research Institute Of Michigan /ID# 273051, Clinton Township, Michigan
  - AA Medical Research Center - Grand Blanc /ID# 253028, Grand Blanc, Michigan
  - June DO, PC /ID# 253030, Lansing, Michigan
  - Kansas City Physician Partners /ID# 254786, Kansas City, Missouri
  - Logan Health Research - Glacier View Research Institute - Rheumatology /ID# 252808, Kalispell, Montana
  - Dartmouth-Hitchcock Medical Center /ID# 254923, Lebanon, New Hampshire
  - Arthritis and Osteoporosis Associates of New Mexico /ID# 252818, Las Cruces, New Mexico
  - Inspire Santa Fe Medical Group /ID# 275947, Santa Fe, New Mexico
  - Joseph S. and Diane H. Steinberg Ambulatory Care Center /ID# 253592, Brooklyn, New York
  - NYU Langone Orthopedic Center /ID# 253613, New York, New York
  - St. Lawrence Health System /ID# 253598, Potsdam, New York
  - Urban Health Plan /ID# 268059, The Bronx, New York
  - Joint And Muscle Research Institute /ID# 272845, Charlotte, North Carolina
  - DJL Clinical Research, PLLC /ID# 253620, Charlotte, North Carolina
  - Raleigh Medical Group /ID# 256328, Raleigh, North Carolina
  - Accellacare - Salisbury /ID# 253608, Salisbury, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 254125, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center /ID# 259174, Cincinnati, Ohio
  - Paramount Medical Research and Consulting /ID# 253016, Middleburg Heights, Ohio
  - Clinical Research Source, Inc. /ID# 253027, Perrysburg, Ohio
  - Oklahoma Medical Research Foundation /ID# 263509, Oklahoma City, Oklahoma
  - Rheumatology Associates of Oklahoma /ID# 253012, Oklahoma City, Oklahoma
  - Clinical Research of Philadelphia, LLC /ID# 254156, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center /ID# 256661, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center /ID# 263686, Pittsburgh, Pennsylvania
  - Low Country Rheumatology /ID# 272956, Summerville, South Carolina
  - West Tennessee Research Institute /ID# 252807, Jackson, Tennessee
  - Shelby Research /ID# 256937, Memphis, Tennessee
  - Arthritis and Rheumatology Research Institute, PLLC /ID# 253014, Allen, Texas
  - Rheumatology Associates /ID# 276066, Arlington, Texas
  - Arthritis Care of Texas /ID# 261719, Corpus Christi, Texas
  - Texas Arthritis Center /ID# 277049, El Paso, Texas
  - JPS Rheumatology Clinic /ID# 253185, Fort Worth, Texas
  - Arthiritis and Rheumatology Specialists PA /ID# 255950, Fort Worth, Texas
  - Integrative Rheumatology of South Texas - Harlingen /ID# 261977, Harlingen, Texas
  - Accurate Clinical Research - Houston /ID# 276220, Houston, Texas
  - Accurate Clinical Research Katy /ID# 276459, Katy, Texas
  - R & H Clinical Research - 777 Katy /ID# 254126, Katy, Texas
  - Biopharma Informatic /ID# 273651, Katy, Texas
  - Valley Arthritis Center /ID# 253022, McAllen, Texas
  - Texas Rheumatology Research Institute Llc /Id# 253013, Plano, Texas
  - Epic Medical Research /ID# 255326, Red Oak, Texas
  - Sun Research Institute /ID# 255832, San Antonio, Texas
  - Clinical Trials of Texas, Inc /ID# 254949, San Antonio, Texas
  - Epic Medical Research- San Marcos /ID# 278360, San Marcos, Texas
  - Fort Bend Rheumatology Associates, PLLC /ID# 268492, Sugar Land, Texas
  - DM Clinical Research - Tomball /ID# 255134, Tomball, Texas
  - Carilion Clinic /ID# 253374, Roanoke, Virginia
  - Rheumatology & Pulmonary Clinic /ID# 273561, Beckley, West Virginia
  - Wisconsin Medical Center /ID# 256660, Milwaukee, Wisconsin
- Argentina (10):
  - Fundación Sanatorio Guemes /ID# 254283, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich /ID# 254278, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Italiano La Plata /ID# 254284, La Plata, Buenos Aires
  - CER Instituto Medico /ID# 255302, Quilmes, Buenos Aires
  - Organizacion Medica de Investigacion (OMI) /ID# 254281, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Fundacion CIDEA /ID# 254279, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto Medico Especializado /ID# 255281, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Aprillus Asistencia e Investigacion /ID# 254276, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto CAICI S.R.L /ID# 254280, Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas Tucuman /ID# 254274, San Miguel de Tucumán, Tucumán Province
- Australia (8):
  - Emeritus Research Sydney /ID# 256249, Botany, New South Wales
  - Concord Repatriation General Hospital /ID# 257945, Concord, New South Wales
  - Momentum Clinical Research /ID# 253542, Darlinghurst, New South Wales
  - Royal Darwin Hospital /ID# 263160, Tiwi, Northern Territory
  - The Queen Elizabeth Hospital /ID# 253826, Woodville, South Australia
  - Emeritus Research /ID# 256800, Camberwell, Victoria
  - Monash Health - Monash Medical Centre /ID# 255678, Clayton, Victoria
  - Colin Bayliss Research and Teaching Unit /ID# 261077, Victoria Park, Western Australia
- Belgium (3):
  - ZAS Palfijn /ID# 252802, Merksem, Antwerpen
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 261997, Anderlecht, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 269065, Jette, Brussels Capital
- Bosnia and Herzegovina (5):
  - Institute of Physical Medicine,Rehab. and Orthopedic Surgery Dr.Miroslav Zotovic /ID# 262588, Banja Luka, Republika Srpska
  - Klinicki centar Banja Luka /ID# 253581, Banja Luka, Republika Srpska
  - Klinicki centar Banja Luka /ID# 253582, Banja Luka, Republika Srpska
  - Clinical Center University of Sarajevo /ID# 253583, Sarajevo
  - Polyclinic Srce Sarajeva /ID# 255475, Sarajevo
- Brazil (9):
  - CEDOES - Centro de Diagnóstico e Pesquisa da Osteoporose do Espírito Santo /ID# 254588, Vitória, Espírito Santo
  - SER - Servicos Especializados em Reumatologia da Bahia /ID# 253354, Salvador, Estado de Bahia
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 253346, Juiz de Fora, Minas Gerais
  - Nossa Saude Pesquisa Ltda. /ID# 253274, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 253357, Porto Alegre, Rio Grande do Sul
  - LMK Sevicos Medicos S/S /ID# 253353, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto /ID# 261024, São José do Rio Preto, São Paulo
  - Hospital do Rim /ID# 253983, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 254316, São Paulo
- Bulgaria (9):
  - Mc Excelsior /ID# 272499, Sofiya, Sofia
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 252642, Sofiya, Sofia
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 252643, Sofiya, Sofia
  - Umbal Kaspela /ID# 252645, Plovdiv
  - Medical Center Artmed Ltd /Id# 254572, Plovdiv
  - Medical center Unimed /ID# 253324, Plovdiv
  - Medical center Teodora /ID# 252646, Rousse
  - Military Medical Academy Multiprofile Hospital /ID# 252644, Sofia
  - Medical Center Academy /ID# 253322, Sofia
- Canada (5):
  - University of Calgary /ID# 259515, Calgary, Alberta
  - University of Alberta Hospital /ID# 259516, Edmonton, Alberta
  - University of Manitoba /ID# 259517, Winnipeg, Manitoba
  - Toronto Western Hospital /ID# 254017, Toronto, Ontario
  - CIUSSS de l'Estrie - CHUS /ID# 254716, Sherbrooke, Quebec
- Chile (5):
  - Hospital Guillermo Grant Benavente de Concepción /ID# 254841, Concepción, Bio-Bio
  - Centro Internacional de Estudios Clinicos - CIEC /ID# 254838, Santiago, Region Metropolitana Santiago
  - Servicio de Salud Araucanía Norte Hospital Victoria /ID# 255179, Victoria, Región de la Araucanía
  - Inmunocel /Id# 256390, Las Condes, Santiago Metropolitan
  - Investigaciones Medicas Limitada /Id# 254842, Providencia
- China (40):
  - The first affiliated hospital of bengbu medical college /ID# 252853, Bengbu, Anhui
  - China-Japan Friendship Hospital /ID# 253048, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 253138, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 253045, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University /ID# 252630, Xiamen, Fujian
  - Guangdong Provincial Peoples Hospital /ID# 252920, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University /ID# 252921, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University /ID# 253137, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical University /ID# 252927, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University /ID# 252923, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College /ID# 253426, Shantou, Guangdong
  - The First Affiliated Hospital Of Guangxi Medical University /ID# 272798, Nanning, Guangxi
  - The First Affiliated Hospital Of Henan University Of Science &Technology /ID# 272929, Luoyang, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 252963, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 252632, Wuhan, Hubei
  - Zhuzhou Central Hospital /ID# 252962, Zhuzhou, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University /ID# 252629, Hohhot, Inner Mongolia
  - The First People's Hospital of Changzhou /ID# 252992, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital /ID# 253042, Nanjing, Jiangsu
  - Affiliated hospital of nantong university /ID# 252991, Nantong, Jiangsu
  - Wuxi People's Hospital /ID# 253858, Wuxi, Jiangsu
  - Xuzhou Central Hospital /ID# 252922, Xuzhou, Jiangsu
  - Yancheng First People's Hospital /ID# 254599, Yancheng, Jiangsu
  - Northern Jiangsu People's Hospital /ID# 252945, Yangzhou, Jiangsu
  - The First People's Hospital of Jiujiang /ID# 252989, Jiujiang, Jiangxi
  - Jiangxi Provincial People's Hospital /ID# 252940, Nanchang, Jiangxi
  - Jiangxi Pingxiang Peoples Hospital /ID# 252919, Pingxiang, Jiangxi
  - The First Hospital of Jilin University /ID# 252771, Changchun, Jilin
  - Second Affiliated Hospital of Xian Jiaotong University /ID# 252861, Xi'an, Shaanxi
  - Jining No.1 People's Hospital /ID# 252897, Jining, Shandong
  - Linyi People's Hospital /ID# 252898, Linyi, Shandong
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 263435, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 252854, Chengdu, Sichuan
  - Mianyang Central Hospital /ID# 272850, Mianyang, Sichuan
  - Tianjin Medical University General Hospital /ID# 252868, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region /ID# 266897, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University /ID# 252925, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 252633, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital /ID# 253860, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 253649, Wenzhou, Zhejiang
- Colombia (6):
  - IPS Suramericana SAS - IPS Sura San Diego /ID# 261536, Medellín, Antioquia
  - Hospital Pablo Tobón Uribe /ID# 254101, Medellín, Antioquia
  - Centro de Investigacion en Reumatologia y especialidades Medicas S.A.S- CIREEM /ID# 254097, Bogotá, Cundinamarca
  - Healthy Medical Center S.A.S /ID# 254098, Zipaquirá, Cundinamarca
  - Fundacion Oftalmologica de Santander - FOSCAL /ID# 254100, Bucaramanga, Santander Department
  - Clinica de la Costa S.A.S /ID# 260727, Barranquilla
- Croatia (6):
  - Poliklinika Bonifarm /ID# 252846, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 252965, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek /ID# 252847, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Rijeka /ID# 252848, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 252849, Split, Split-Dalmatia County
  - Opća Bolnica Zadar /ID# 272415, Zadar, Zadar County
- Estonia (4):
  - Innomedica /ID# 253722, Tallinn, Harju
  - East Tallinn Central Hospital - Magdaleena Unit /ID# 253721, Tallinn, Harju
  - North Estonia Medical Centre Foundation /ID# 253723, Tallinn, Harju
  - MediTrials /ID# 253720, Tartu, Tartu
- France (3):
  - CHU Toulouse - Hopital Rangueil /ID# 254148, Toulouse, Haute-Garonne
  - HCL - Hopital de la Croix-Rousse /ID# 254147, Lyon, Rhone
  - Hopital Pitie Salpetriere /ID# 253009, Paris, Île-de-France Region
- Germany (5):
  - Krankenhaus Porz am Rhein /ID# 254373, Cologne, North Rhine-Westphalia
  - Universitaetsmedizin Mainz /ID# 260735, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 270832, Dresden, Saxony
  - Immanuel Krankenhaus Berlin /ID# 253389, Buch
  - Fraunhofer Institute for Translational Medicine & Pharmacology ITMP /ID# 253734, Frankfurt am Main
- Greece (3):
  - General Hospital of Athens Laiko /ID# 252952, Athens, Attica
  - University General Hospital Attikon /ID# 253209, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 252951, Heraklion, Crete
- Guatemala (4):
  - Clinica Medica Especializada en Medicina Interna y Reumatologia /ID# 261156, Guatemala City
  - Clinica Medica Reumatologica /ID# 255009, Guatemala City
  - Clinica Especializada en Medicina Interna /ID# 255006, Guatemala City
  - Clínica Médica Especializada en Medicina Interna y Reumatologia /ID# 257248, Guatemala City
- Hungary (5):
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 254552, Pécs, Baranya
  - Vital-Medicina Kft. /ID# 252876, Veszprém, Fejér
  - Debreceni Egyetem-Klinikai Kozpont /ID# 252877, Debrecen, Hajdú-Bihar
  - Vita Verum Medical Bt. /ID# 273579, Székesfehérvár, Szekesfehervar
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz /ID# 252886, Gyula
- Israel (6):
  - Meir Medical Center /ID# 254187, Kfar Saba, Central District
  - Hadassah Medical Center-Hebrew University /ID# 252654, Jerusalem, Jerusalem
  - Galilee Medical Center /ID# 252859, Nahariya, Northern District
  - The Chaim Sheba Medical Center /ID# 252857, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 252858, Tel Aviv, Tel Aviv
  - The Lady Davis Carmel Medical Center /ID# 253303, Haifa
- Italy (5):
  - Azienda Ospedaliera San Camillo Forlanini /ID# 253680, Rome, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 254288, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 254138, Ancona
  - Azienda Ospedale-Universita Padova /ID# 253704, Padua
  - Azienda Ospedaliero Universitaria Pisana /ID# 254289, Pisa
- Japan (11):
  - Hospital Of The University Of Occupational And Environmental Health, Japan /ID# 253269, Kitakyushu-shi, Fukuoka
  - Hokkaido University Hospital /ID# 253306, Sapporo, Hokkaido
  - Tohoku University Hospital /ID# 253267, Sendai, Miyagi
  - University of Miyazaki Hospital /ID# 253416, Miyazaki, Miyazaki
  - Okayama University Hospital /ID# 253821, Okayama, Okayama-ken
  - Shinkenko Clinic /ID# 253271, Naha, Okinawa
  - Saitama Medical Center /ID# 253263, Kawagoe, Saitama
  - Institute of Science Tokyo Hospital /ID# 254430, Bunkyo-ku, Tokyo
  - University of Yamanashi Hospital /ID# 253264, Chuo-shi, Yamanashi
  - National Hospital Org Chiba Medical Center Chibahigashi National Hospital /ID# 253268, Chiba
  - Hiroshima University Hospital /ID# 273658, Hiroshima
- Latvia (5):
  - Riga East Clinical University Hospital /ID# 253751, Riga, Rīga
  - M & M Centrs LTD /ID# 253752, Ādaži
  - Daugavpils Regional Hospital /ID# 253754, Daugavpils
  - Dr. Saulites-Kandevicas PP in Cardiology and Rheumatology /ID# 273246, Liepāja
  - Pauls Stradins Clinical University Hospital /ID# 253750, Riga
- Lithuania (5):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 253755, Kaunas
  - Republic Klaipeda Hospital /ID# 253759, Klaipėda
  - Klaipeda University Hospital, Klaipeda Hospital /ID# 253757, Klaipėda
  - Inlita - Santara KTC /ID# 253758, Vilnius
  - Vilnius University Hospital Santaros Klinikos /ID# 253756, Vilnius
- Mexico (7):
  - Centro de Investigacion Medica Dr. Alberto Bazzoni CIMAB S.A de C.V. /ID# 261462, Torreón, Coahuila
  - Morales Vargas Centro de Investigacion S.C. /ID# 254661, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 253966, Guadalajara, Jalisco
  - Grupo Clinico Catei Sociedad Civil /Id# 257700, Guadalajara, Jalisco
  - Hospital de Jesus /ID# 255146, Mexico City, Mexico City
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 253965, Mexico City, Mexico City
  - Medical Care & Research SA de CV /ID# 260825, Mérida, Yucatán
- New Zealand (2):
  - Aotearoa Clinical Trials /ID# 253555, Papatoetoe, Auckland
  - North Shore Hospital /ID# 253554, Takapuna, Auckland
- Poland (5):
  - Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im. Wiktora Degi /ID# 252964, Poznan, Greater Poland Voivodeship
  - MICS Centrum Medyczne Bydgoszcz /ID# 253281, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela /ID# 253233, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Warszawa /ID# 253273, Warsaw, Masovian Voivodeship
  - ETYKA-Osrodek Badan Klinicznych /ID# 252967, Olsztyn, Warmian-Masurian Voivodeship
- Portugal (4):
  - Centro Hospitalar do Tamega e Sousa - Hospital Padre Americo /ID# 252911, Guilhufe, Porto District
  - Hospital Garcia de Orta /ID# 252903, Almada, Setúbal District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 252902, Ponte de Lima, Viana do Castelo District
  - Centro Hospitalar Universitario do Porto, EPE - Hospital Santo Antonio /ID# 252899, Porto
- Puerto Rico (5):
  - Clinical Research Investigator Group, LLC /ID# 259170, Bayamón
  - Clinical Research Puerto Rico /ID# 256352, San Juan
  - GCM Medical Group PSC /ID# 253039, San Juan
  - Caribbean Medical Research Center /ID# 254882, San Juan
  - Mindful Medical Research /ID# 253040, San Juan
- Romania (3):
  - Spitalul Clinic Judetean de Urgenta Cluj -Napoca /ID# 252904, Cluj-Napoca, Cluj
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL /ID# 253207, Brasov
  - Spitalul Clinic Sf. Maria /ID# 252905, Bucharest
- Serbia (8):
  - Institute for Rheumatology /ID# 253172, Belgrade, Beograd
  - Institute for Rheumatology /ID# 253173, Belgrade, Beograd
  - Institute for Rheumatology /ID# 253174, Belgrade, Beograd
  - Institute for Rheumatology /ID# 253175, Belgrade, Beograd
  - Military Medical Academy /ID# 264235, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 253179, Belgrade, Beograd
  - General Hospital Djordje Joanovic /ID# 253177, Zrenjanin, Vojvodina
  - University Clinical Center Vojvodina /ID# 253176, Novi Sad
- Slovakia (5):
  - ARTROMAC n.o. /ID# 253056, Košice, Košice Region
  - Narodny Ustav Reumatickych Chorob Piestany /ID# 273341, Piešťany, Trnava Region
  - ZAZABIE s. r .o. /ID# 255793, Košice II
  - Thermium s.r.o. /ID# 260839, Piešťany
  - MEDMAN s.r.o. /ID# 252950, Martin, Žilina Region
- South Africa (7):
  - Wits Clinical Research /ID# 252931, Johannesburg, Gauteng
  - University of Pretoria /ID# 252932, Pretoria, Gauteng
  - Dr Elsa van Duuren /ID# 254218, Pretoria, Gauteng
  - Dr Asokan Naidoo /ID# 253351, Umhlanga, KwaZulu-Natal
  - Winelands Medical Research - Somerset West /ID# 254614, Cape Town, Western Cape
  - Arthritis Clinical Research Trials /ID# 253349, Cape Town, Western Cape
  - Winelands Medical Research Centre /ID# 252934, Stellenbosch, Western Cape
- South Korea (5):
  - SoonChunHyang University Hospital Cheonan /ID# 254777, Cheonan-si, Chungcheongnam-do
  - Chonnam National University Bitgoeul Hospital /ID# 254675, Gwangju, Gwangju Gwang Yeogsi
  - Hanyang University Seoul Hospital /ID# 252955, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 254022, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 252958, Seoul, Seoul Teugbyeolsi
- Spain (3):
  - Complejo Hospitalario Universitario A Coruña /ID# 253123, A Coruña, A Coruna
  - Hospital Meixoeiro (CHUVI) /ID# 253124, Vigo, Pontevedra
  - Hospital Universitario Virgen de Valme /ID# 253121, Seville
- Switzerland (3):
  - University Hospital Basel /ID# 252907, Basel Town, Canton of Basel-City
  - Kantonsspital St. Gallen /ID# 252906, Sankt Gallen, Canton of St. Gallen
  - Inselspital, Universitaetsspital Bern /ID# 252909, Bern
- Taiwan (3):
  - National Taiwan University Hospital /ID# 252937, Taipei City, Taipei
  - Chang Gung Mem Hosp Keelung /ID# 253636, Keelung
  - China Medical University Hospital /ID# 252936, Taichung
- Turkey (Türkiye) (8):
  - Hacettepe Universitesi Tip Fak /ID# 253266, Sihhiye, Ankara, Ankara
  - Gazi Universitesi Tip Fakultes /ID# 252843, Yenimahalle, Ankara
  - Sanko Universitesi Hastanesi /ID# 252841, Şehitkamil, Gaziantep
  - Akdeniz Universitesi Tip Fakul /ID# 252839, Antalya
  - Basaksehir Cam ve Sakura Sehir Hastanesi /ID# 253557, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 252844, Istanbul
  - Necmettin Erbakan Universitesi /ID# 252837, Meram Konya
  - Karadeniz Technical University Farabi Hospital /ID# 252845, Trabzon
- United Kingdom (7):
  - North West Anglia NHS Foundation Trust /ID# 254590, Bretton, Cambridgeshire
  - Guy's Hospital /ID# 252978, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 252982, Southampton, Hampshire
  - Northampton General Hospital NHS Trust /ID# 254813, Northampton, Northamptonshire
  - Western Health and Social Care Trust /ID# 254592, Londonderry, Northern Ireland
  - Luton and Dunstable Hospital NHS Foundation Trust /ID# 255323, Luton
  - Portsmouth Hospitals University NHS Trust /ID# 252986, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-699